CLINICAL TRIAL: NCT04445662
Title: Financial Incentives for Homeless Smokers: A Community-based RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Travis Paul Baggett, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000034; R01CA235617-01 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Smoking
Keywords: Smoking Cessation; Homelessness; Financial Incentives
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (n=90) (Active Comparator): * Varenicline
  * Tobacco coaching
  * Saliva cotinine monitoring with fixed payments ($10) regardless of results
  Interventions: Drug: Varenicline; Behavioral: Tobacco coaching
- Financial incentives (n=90) (Experimental): * Varenicline
  * Tobacco coaching
  * Saliva cotinine monitoring with escalating payments ($25-70) for levels <30 ng/ml
  Interventions: Behavioral: Financial incentives; Drug: Varenicline; Behavioral: Tobacco coaching

INTERVENTIONS:
Behavioral: Financial incentives — Escalating financial rewards for saliva cotinine levels <30 ng/mL, assessed 10 times over 12 weeks
  Other Names: Contingency management
  Arms: Financial incentives (n=90)
Drug: Varenicline — * Day 1 - 3: 0.5 mg daily
  * Day 4 - 7: 0.5 mg twice daily
  * Day 8 - Week 12: 1 mg twice daily
  * Dose/schedule may be adjusted based on medical history and clinician judgement
  Other Names: Chantix
Behavioral: Tobacco coaching — 5 one-on-one tobacco cessation coaching sessions over 12 weeks
  Other Names: Smoking cessation counseling

SUMMARY:
This community-based randomized controlled trial will test the effect of contingent financial rewards on smoking abstinence among homeless-experienced adult cigarette smokers. Participants will be recruited from 3 Boston Health Care for the Homeless Program locations: a shelter clinic, a day center clinic, and a medical center clinic. All participants will be offered a varenicline prescription and tobacco coaching. Incentive arm participants will receive escalating financial rewards for saliva cotinine levels <30 ng/ml, assessed 10 times over 12 weeks. Embedded qualitative interviews will explore the mechanisms of on-treatment and post-treatment effects of financial incentives on smoking abstinence in the context of homelessness.

DETAILED DESCRIPTION:
People experiencing homelessness have a 3.5-fold higher prevalence of cigarette smoking in comparison to non-homeless people, contributing to 2-fold higher rates of lung cancer and 3- to 5-fold higher rates of tobacco-attributable death. Homeless smokers want to quit, but studies have not yet uncovered the optimal approach to help them do so. In an 8-week pilot randomized controlled trial (RCT) at Boston Health Care for the Homeless Program (BHCHP), we found that financial incentives for smoking abstinence were associated with 7-fold higher odds of brief smoking abstinence in comparison to a non-incentivized control condition. These results suggest that financial incentives are a promising approach for reducing smoking in this vulnerable population, but further investigation in a larger sample is needed to improve the duration of on-treatment abstinence, assess post-treatment effects, and better understand mechanisms of action and contextual factors that may influence treatment response.

To address the above gaps in evidence, we will conduct a community-based RCT of financial incentives for smoking abstinence among adult smokers at BHCHP. Recognized as a leader in homeless health care, BHCHP serves 12,000 currently and formerly homeless patients annually throughout greater Boston. We will randomize 180 participants recruited from 3 BHCHP sites: a shelter clinic, a day center clinic, and a medical center clinic. All participants will be offered 12 weeks of varenicline, 5 sessions of tobacco coaching, and 10 cotinine monitoring visits over a 12-week period. Participants randomized to the financial incentives arm (n=90) will receive escalating debit card payments (range $25-$70) at each monitoring visit for saliva cotinine levels <30 ng/ml. Control arm participants (n=90) will receive a fixed payment ($10) at each monitoring visit regardless of their saliva cotinine level. We will use an embedded-experiment mixed methods design, where qualitative ('qual') data collection is embedded within a larger quantitative ('QUAN') RCT with the following specific aims:

Aim 1. (QUAN) To determine the effect of the financial incentives intervention on cotinine-verified 7-day smoking abstinence at A) the end of treatment (12 weeks) and B) 12 weeks after treatment (24 weeks).

Hypotheses: Incentive arm participants will have significantly greater cotinine-verified 7-day smoking abstinence than control arm participants at A) 12 weeks and B) 24 weeks.

Aim 2. (qual) To assess why, how, and under what circumstances homeless smokers A) achieve abstinence in response to financial incentives and B) maintain abstinence after incentives are stopped.

Interviews with participants at A) 12 weeks (N=30) and B) 24 weeks (N=20) will examine cognitive ('why?'), procedural ('how?'), and contextual ('under what circumstances?') dimensions of their response to financial incentives to generate hypotheses about potential mechanisms for on-treatment and post-treatment effects and to inform modifications of the intervention for future use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Lifetime smoker of ≥100 cigarettes with current daily smoking of ≥5 cigarettes per day, verified by a saliva cotinine level of ≥30 ng/mL
* Ready to try quitting smoking within the next 3 months
* Proficient in English
* Currently or formerly homeless
* Have a primary care provider within BHCHP system

Exclusion Criteria:

* Unable to provide informed consent
* History of allergic reaction to varenicline
* Currently pregnant, planning to become pregnant, or breastfeeding
* Past-month suicidal ideation with plan or intent, or past 12-month history of suicidal behaviors or attempts
* Psychiatric hospitalization in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis Baggett, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Boston Health Care for the Homeless Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data and personal health information involved, we do not plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between 2021-2024 at Boston Health Care for the Homeless Program (BHCHP), a federally funded Health Care for the Homeless (HCH) organization. Participants were recruited via in-person outreach at BHCHP clinic sites, telephone outreach to BHCHP patients with a past-year clinical encounter and electronic health record (EHR) documentation of current smoking, self-referrals in response to flyers or word of mouth, and referrals from BHCHP clinicians.
Pre-assignment Details: Enrolled participants provided written informed consent and completed a staff-administered baseline survey. To be assigned a study arm, enrolled participants were asked to attend a randomization appointment within 4 weeks of enrollment.
Groups:
- Control (n=69): * Varenicline
  * Tobacco coaching
  * Saliva cotinine monitoring with fixed payments ($10) regardless of results
  Varenicline: - Day 1 - 3: 0.5 mg daily
  * Day 4 - 7: 0.5 mg twice daily
  * Day 8 - Week 12: 1 mg twice daily
  * Dose/schedule may be adjusted based on medical history and clinician judgement
  Tobacco coaching: 5 one-on-one tobacco cessation coaching sessions over 12 weeks
- Financial incentives (n=69): * Varenicline
  * Tobacco coaching
  * Saliva cotinine monitoring with escalating payments ($25-70) for levels <30 ng/ml
  Financial incentives: Escalating financial rewards for saliva cotinine levels <30 ng/mL, assessed 10 times over 12 weeks
  Varenicline: - Day 1 - 3: 0.5 mg daily
  * Day 4 - 7: 0.5 mg twice daily
  * Day 8 - Week 12: 1 mg twice daily
  * Dose/schedule may be adjusted based on medical history and clinician judgement
  Tobacco coaching: 5 one-on-one tobacco cessation coaching sessions over 12 weeks
Period: On treatment (0-12 weeks)
Arm/Group | Control (n=69) | Financial incentives (n=69)
Started | 69 | 69
Completed | 65 | 64
Not Completed | 4 | 5
Not completed — Deemed ineligible after randomization due to non-smoking status | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Withdrawn by PI due to behavioral concerns | 1 | 0
Period: Post-treatment (12-24 weeks)
Arm/Group | Control (n=69) | Financial incentives (n=69)
Started | 65 | 64
Completed | 64 | 64
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control (n=68): * Varenicline
  * Tobacco coaching
  * Saliva cotinine monitoring with fixed payments ($10) regardless of results
  Varenicline: - Day 1 - 3: 0.5 mg daily
  * Day 4 - 7: 0.5 mg twice daily
  * Day 8 - Week 12: 1 mg twice daily
  * Dose/schedule may be adjusted based on medical history and clinician judgement
  Tobacco coaching: 5 one-on-one tobacco cessation coaching sessions over 12 weeks
- Total: Total of all reporting groups
Arm/Group | Control (n=68) | Financial incentives (n=69) | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (10.3) | 49.0 (10.1) | 50.1 (10.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 44 | 56 | 100
  Gender: Female | 24 | 11 | 35
  Gender: Other | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic/Latine | 6 | 17 | 23
  Race/Ethnicity: Non-Hispanic Black | 17 | 14 | 31
  Race/Ethnicity: Non-Hispanic White | 34 | 26 | 60
  Race/Ethnicity: Non-Hispanic Other | 11 | 10 | 21
  Race/Ethnicity: Unknown | 0 | 2 | 2
Homelessness status [Count of Participants; unit: Participants]
  Currently homeless | 36 | 35 | 71
  Formerly homeless | 32 | 34 | 66
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes] — Self-reported number of cigarettes smoked per day at baseline.
  cigarettes | 14.3 (6.8) | 14.1 (7.3) | 14.2 (7.0)
Alcohol use disorder [Count of Participants; unit: Participants] — Based on summed score of >= 8 on the Alcohol Use Disorders Identification Test (AUDIT)
  Participants | 18 | 9 | 27
Drug use disorder [Count of Participants; unit: Participants] — Based on summed score of >= 3 on the Drug Abuse Screening Test (DAST-10) . Population: 1 control arm participant did not answer enough questions to be categorized.
  Participants
    number analyzed (Participants) | 67 | 69 | 136
    (all) | 40 | 39 | 79
Moderate/severe depression [Count of Participants; unit: Participants] — Based on summed score of >= 10 on the PHQ-9.
  Participants | 25 | 27 | 52
Moderate/severe anxiety [Count of Participants; unit: Participants] — Based on summed score of >=10 on the GAD-7. Population: 1 incentives arm participant did not answer enough questions to be categorized.
  Participants
    number analyzed (Participants) | 68 | 68 | 136
    (all) | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Cotinine-verified 7-day Smoking Abstinence at 12 Weeks
Description: Point-prevalent smoking abstinence, defined as self-report of not smoking in the past 7 days and verified by a salivary cotinine level <10 ng/ml.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control (n=68) | Financial incentives (n=69)
Number analyzed (Participants) | 68 | 69
Participants | 3 | 4
Statistical Analysis 1: Comparison: Control (n=68) vs Financial incentives (n=69); Test type: Superiority; p = 0.71, Chi-squared

2. Secondary Outcome: Cotinine-verified 7-day Smoking Abstinence at 24 Weeks
Description: as for outcome 1
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control (n=68) | Financial incentives (n=69)
Number analyzed (Participants) | 68 | 69
Participants | 3 | 5
Statistical Analysis 1: Comparison: Control (n=68) vs Financial incentives (n=69); Test type: Superiority; p = 0.48, Chi-squared

ADVERSE EVENTS:
Time Frame: From enrollment until end of study follow-up at 24 weeks.
Description: Participant were asked whether they had experienced specific symptoms linked with varenicline use (e.g. abnormal dreams, headaches, nausea, vomiting, and suicidality) at each cotinine monitoring visit. Participants could also report adverse events at any other study visit or via phone call to study staff. For each AE reported, study staff assessed date of onset, level of severity, resolution status, expectedness, and relatedness to study protocol.
Arm/Group | Control (n=69) | Financial incentives (n=69)
All-Cause Mortality (participants affected / at risk) | 1/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 3/69 | 2/69
Other Adverse Events (participants affected / at risk) | 43/69 | 37/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (n=69) (N=69) | Financial incentives (n=69) (N=69)
Suicidality (Psychiatric disorders) | 2 (2) | 2 (2) — Severe suicidal thoughts or actions resulting in psychiatric hospitalization.
Collapsed (General disorders) | 1 (1) | 0 (0) — Sudden unconsciousness resulting in hospitalization due to stress and dehydration.
Death (General disorders) | 1 (1) | 0 (0) — Died before end of study follow-up period. Cause unclear but deemed unrelated to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (n=69) (N=69) | Financial incentives (n=69) (N=69)
Headache (General disorders) | 23 (30) | 18 (21)
Abnormal Dreams (Psychiatric disorders) | 22 (24) | 24 (27) — Self-reported unusually vivid or troubling dreams.
Nausea (Gastrointestinal disorders) | 22 (29) | 17 (24)
Insomnia (General disorders) | 19 (20) | 10 (12)
Aggressive/erratic behavior (Psychiatric disorders) | 8 (9) | 8 (8) — Self-reported increase in feelings of aggression or aggressive/erratic behaviors.
Vomiting (Gastrointestinal disorders) | 8 (9) | 7 (9)
Suicidality (Psychiatric disorders) | 4 (4) | 3 (3) — Self-reported suicidal thoughts or behaviors not causing psychiatric hospitalization.

LIMITATIONS AND CAVEATS:
Various limitations led to lower than anticipated enrollment and limited statistical power. The COVID-19 pandemic substantially delayed study launch. Shortly after the initial launch, recruitment was halted and delayed again due to the recall and global shortage of varenicline (the study medication). Reductions in foot traffic at recruitment sites (due to COVID-19 and fluctuating local patterns of and responses to homelessness) led to slower rates of recruitment once the study was relaunched.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT04445662/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04445662/ICF_001.pdf